CLINICAL TRIAL: NCT03130582
Title: 2008 WHO Myeloid and Lymphocytic Tumor Diagnostic Criteria
Brief Title: High-dose Etoposide Could Discriminate Patients With Refractory/Relapsed Lymphoma Benefit From APBSCT
Status: Completed | Type: Observational
Sponsor: Yang Jun (Other)
Responsible Party: Sponsor-Investigator, Yang Jun, Principal Investigator, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Other Study IDs: 2015KY143
Record Dates: First submitted 2017-04-22; First posted 2017-04-26 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Lymphoma
Keywords: high-dose etoposide,autologous peripheral blood stem cell transplantation
MeSH Terms: conditions — Lymphoma | interventions — Etoposide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Disease status at mobilization PR
  Interventions: Drug: high-dose etoposide
- Disease status at mobilization PD
  Interventions: Drug: high-dose etoposide

INTERVENTIONS:
Drug: high-dose etoposide — an epipodophyllotoxin, is one of the most common chemotherapy agents for lymphoma without reciprocal resistance with other kinds of agents.

SUMMARY:
patients with refractory /relapsed lymphoma received high-dose etoposide for hematopoietic stem cell (HSC) mobilization.All patients received high-dose etoposide 20-25 mg/kg/d intravenously for two consecutive days followed by rhG-CSF10ug/kg/day subcutaneously at 48 hours after chemotherapy; rhG-CSF was continued until the end of harvesting for HSCs/HPCs. Peripheral blood counts were performed daily for all patients following the initiating of rhG-CSF. Leukapheresis was performed when peripheral blood white blood count exceeded 4×109/L with blood cell The harvested cells reached at least 2*108/kg for mononuclear cells and/or 2*106/kg for CD34+ cells with once to twice leukapheresis. The final product was kept frozen in liquid nitrogen.Auto-PBSCT

ELIGIBILITY:
Inclusion Criteria:

* relapsed/refractory lymphoma ,siut APBSCT

Exclusion Criteria:

* bone marrow without involvement by lymphoma cells

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients with refractory/relapsed lymphoma
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2005-11 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
death | 10 years
  death
CR | 10 years
  Complete response
relapse | 10 years
  relapse